CLINICAL TRIAL: NCT03815968
Title: The Influence of Low Sodium Diet on an Amniotic Fluid Index in a Patient That Diagnosed With Oligohydramnios and Assigned for Conservative Management - a Randomized Controlled Trial
Brief Title: Low Sodium Diet in Oligohydramnios Assigned for Conservative Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Levy, MD, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0008-19-WOMC
Record Dates: First submitted 2019-01-19; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Oligohydramnios
Keywords: oligohydroamnios; low salt diet
MeSH Terms: conditions — Oligohydramnios | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low sodium diet (Experimental): women diagnosed with oligohydramnios designated for conservative management applying a low-salt diet.
  Interventions: Other: low sodium diet
- regular diet (No Intervention): women diagnosed with oligohydramnios designated for conservative management applying a regular diet.

INTERVENTIONS:
Other: low sodium diet — included in the diet mostly low sodium food. avoid tinned or smoked, food. avoid adding salt to the food.
  Other Names: low salt diet
  Arms: low sodium diet

SUMMARY:
The investigators want to examine whether low salt diet can increase the amniotic fluid index in patients diagnosed with oligohydramnios and assigned for conservative management. A randomized controlled trial

DETAILED DESCRIPTION:
Few studies have addressed the changes in maternal diet as affecting the composition and amount of amniotic fluid.

Some articles have shown an increase in amniotic fluid volume as a result of maternal hydration during pregnancy through intravenous fluid infusions and oral fluid intake, the increase was evident in women with amniotic fluid and women with normal amniotic fluid volume. In a mechanism similar to that of liquid hydration, a low-salt diet may lead to an increase in the volume of amniotic fluid.

The investigators would like to examine whether a low-salt diet in women with amniotic fluid is able to significantly increase the amount of amniotic fluid compared with a regular diet.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24-37 weeks of gestation, single fetus, who were diagnosed with an amniotic fluid index at the 5th percentile or below, according to the current gestational age
* No medical indication for immediate delivery

Exclusion Criteria:

* Refusal to participate in the study
* A medical recommendation for delivery within two weeks of diagnosis
* Fetal malformation or proof of fetal infection that known to cause oligohydramnios (eg CMV).
* Premature rupture of membrane
* Multiple pregnancy
* Medical contraindication to the low-salt diet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
amniotic fluid volume, assessed by ultrasound | two weeks
  amniotic fluid volume after two weeks

SECONDARY OUTCOMES:
gestational age at birth | up to 18 weeks (until delivery)
induction of labor | up to 18 weeks (until delivery)
  The percentage of pregnant women who underwent birth induction
labor type | up to 18 weeks (until delivery)
  Cesarean section, vaginal birth or vaginal birth
Pregnancy and childbirth complications | up to 18 weeks (until delivery)
  obstetrics complications and neonatal complications

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Obstetrics & Gynecology, affiliated with Sackler Faculty of Medicine, Tel Aviv University, Holon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rabie N, Magann E, Steelman S, Ounpraseuth S. Oligohydramnios in complicated and uncomplicated pregnancy: a systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2017 Apr;49(4):442-449. doi: 10.1002/uog.15929. PMID 27062200
- [Result] Rainford M, Adair R, Scialli AR, Ghidini A, Spong CY. Amniotic fluid index in the uncomplicated term pregnancy. Prediction of outcome. J Reprod Med. 2001 Jun;46(6):589-92. PMID 11441685
- [Result] Koski KG, Fergusson MA. Amniotic fluid composition responds to changes in maternal dietary carbohydrate and is related to metabolic status in term fetal rats. J Nutr. 1992 Feb;122(2):385-92. doi: 10.1093/jn/122.2.385. PMID 1732479
- [Result] Gurekian CN, Koski KG. Amniotic fluid amino acid concentrations are modified by maternal dietary glucose, gestational age, and fetal growth in rats. J Nutr. 2005 Sep;135(9):2219-24. doi: 10.1093/jn/135.9.2219. PMID 16140901
- [Result] Flack NJ, Sepulveda W, Bower S, Fisk NM. Acute maternal hydration in third-trimester oligohydramnios: effects on amniotic fluid volume, uteroplacental perfusion, and fetal blood flow and urine output. Am J Obstet Gynecol. 1995 Oct;173(4):1186-91. doi: 10.1016/0002-9378(95)91350-5. PMID 7485317
- [Result] Doi S, Osada H, Seki K, Sekiya S. Effect of maternal hydration on oligohydramnios: a comparison of three volume expansion methods. Obstet Gynecol. 1998 Oct;92(4 Pt 1):525-9. doi: 10.1016/s0029-7844(98)00242-7. PMID 9764623
- [Result] Umber A, Chohan MA. Intravenous maternal hydration in third trimester oligohydramnios: effect on amniotic fluid volume. J Coll Physicians Surg Pak. 2007 Jun;17(6):336-9. PMID 17623581
- [Result] Rakova N, Muller DN, Staff AC, Luft FC, Dechend R. Novel ideas about salt, blood pressure, and pregnancy. J Reprod Immunol. 2014 Mar;101-102:135-139. doi: 10.1016/j.jri.2013.04.001. Epub 2013 May 30. PMID 23726817
- [Result] Kirksey A, Pike RL, Callahan JA. Some effects of high and low sodium intakes during pregnancy in the rat. II. Electrolyte concentrations of maternal plasma, muscle, bone and brain and of placenta, amniotic fluid, fetal plasma and total fetus in normal pregnancy. J Nutr. 1962 May;77(1):43-51. doi: 10.1093/jn/77.1.43. No abstract available. PMID 14456322
- [Result] Moore TR, Cayle JE. The amniotic fluid index in normal human pregnancy. Am J Obstet Gynecol. 1990 May;162(5):1168-73. doi: 10.1016/0002-9378(90)90009-v. PMID 2187347